CLINICAL TRIAL: NCT02599038
Title: Serine Supplementation in Nonalcoholic Fatty Liver Disease
Brief Title: Serine Supplementation for Obese Subjects With Fatty Liver Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanns-Ulrich Marschall (Other)
Responsible Party: Sponsor-Investigator, Hanns-Ulrich Marschall, Professor of Clinical Hepatology, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Serine-NAFLD
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; Serine; Glutathione
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Serine supplementation (Experimental): Serine oral administration 20mg/kg/day
  Interventions: Dietary Supplement: Serine supplementation

INTERVENTIONS:
Dietary Supplement: Serine supplementation — Serine supplementation (200 mg/kg/day)

SUMMARY:
In this study, the investigators aim to increase the liver tissue level of GSH in NAFLD patients by short-term dietary serine supplementation and improve their liver function by lowering the oxidative stress resulting from hepatic steatosis.

DETAILED DESCRIPTION:
There is a strong correlation between major adverse health consequences of obesity and development of non-alcoholic fatty liver disease (NAFLD). NAFLD is characterized by abnormal hepatic accumulation of triglycerides and other lipids. It has become a worldwide health problem that accelerates cirrhosis, type 2 diabetes mellitus (T2DM), and especially premature cardiovascular morbidity and mortality.

The plasma level of glutathione (GSH) is typically depleted in individuals with metabolism related disorders. However, cellular GSH levels cannot be increased by supplementing GSH and it must be synthesized within the liver either de novo or by salvation pathway. The investigators found that the level of GSH is not enough to maintain and regulate the thiol redox status of the liver in subjects with high hepatic steatosis at fasting stage due to the depletion of glycine. Glycine can be synthesized via the interconversion of serine through serine hydroxymethyl transferases (SHMT1 and SHMT2) with concomitant conversion of tetrahydrofolate (THF) into 5,10-methylene-THF (CH2-THF). It has been shown that the serine synthesis is downregulated in patients with NAFLD and supplementation of serine has attenuated alcoholic fatty liver by enhancing homocysteine metabolism in mice and rats.

In this study, the investigators aim to increase the liver tissue level of GSH in NAFLD patients by short-term dietary serine supplementation and improve their liver function by lowering the oxidative stress resulting from hepatic steatosis.

Ten obese patients (BMI 30 - 39.9 kg/m2) with ultrasound and CT-verified non-alcoholic fatty liver disease (NAFLD). Subjects will be recruited from the Swedish CArdioPulmonary bioImage Study (SCAPIS) in Gothenburg. The participants in this study (50-65-year-old men and women) are randomly recruited from the Swedish Population and Address Register. Currently, 1050 subjects have been analyzed and 5000 additional subjects will be analyzed over the next 2 years. By January 2015, over 2000 subjects have been analyzed. Each subject is extensively phenotyped over two days. This includes extensive blood samples, anthropometry, carotid and liver ultrasound, and a CT examination that includes coronary calcium score, CT angiography of coronary arteries, thoracic aorta, and assessment of epicardial fat, liver fat, and subcutaneous abdominal fat.

Preliminary analysis of the first 1050 subjects indicates that approximately 20% fulfill the criteria for NAFLD, consistent with data in other western populations.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 - 39.9 kg/m2; stable weight (+/- 2 kg) within the last six months
* Sex Males, pre-, and post-menopausal females
* Women of childbearing potential can only be included if a safe and reliable contraception is used, e.g., oral contraceptives
* Diagnosis NAFLD established by both liver CT and ultrasound
* Consent Patients should have given their written consent to participate in this study

Exclusion Criteria:

* Chronic liver disease other than NAFLD (viral hepatitis, autoimmune liver disease, hemochromatosis, homozygous alpha1-antitrypsin deficiency and Wilson disease)
* Previous gastric or small bowel surgery
* Inflammatory bowel disease
* Uncontrolled diabetes mellitus (fasting blood glucose >6.7 mmol/L), hypothyroidism or hyperthyroidism, or other significant endocrine disease. (A subject who is euthyroid on a stable replacement dose of thyroid hormone is acceptable provided the TSH is within normal range).
* Pregnancy. A urine pregnancy test will be performed the day before start of medication. Women of childbearing potential can only be included if a safe and reliable contraception is used, e.g., oral contraceptives.
* Elevations of transaminases (ALAT/ASAT) or alkaline phosphatase or bilirubin above 2xULN (upper limit of normal) the day before start of serine supplementation.
* Other serious disease, including depressive disorders treated by medication
* Patients who will not comply with the protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Liver fat content | 2 weeks
  Liver fat measured by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Triglycerides | 2 weeks
Cholesterol fractions | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Ulrich Marschall, MD, PhD, Principal Investigator — Sahlgrenska Academy and University Hospital
Locations (2):
- Sweden (2):
  - Hanns-Ulrich Marschall, Gothenburg
  - Sahlgrenska Academy, Gothenburg

IPD SHARING:
Plan to Share IPD: No